CLINICAL TRIAL: NCT00730158
Title: A Phase II Multicenter, Randomized, Placebo Controlled, Double Blinded Clinical Study of KD018 as a Modulator of Irinotecan Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edward Chu, MD (Other)
Collaborators: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor-Investigator, Edward Chu, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-005; ACS IRG 58-012-49
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): irinotecan+ KD018
  Interventions: Drug: KD018; Drug: Irinotecan
- Arm B (Experimental): irinotecan + placebo
  Interventions: Drug: Irinotecan; Drug: Placebo

INTERVENTIONS:
Drug: KD018 — Traditional Chinese Medicine formulation administered orally twice a day for 4 days on days 1-4 every 2 weeks from the second cycle, at a dose of 1,800 mg, twice a day.
  Arms: Arm A
Drug: Irinotecan — Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
  Other Names: Camptosar; CPT-11
Drug: Placebo — Placebo capsules will be administered orally twice a day for 4 days on days 1-4 every 2 weeks.
  Arms: Arm B

SUMMARY:
The proposed plan will investigate the mechanism and efficacy of Chinese herbal medicine as an adjunct to chemotherapy in treatment of patients with metastatic colorectal cancer. Our rationale for the therapeutic use of KD018 is its potential activity in reducing chemotherapy-induced toxicity, especially diarrhea.

DETAILED DESCRIPTION:
KD018 is an oral form of a spray dried aqueous extract composed of four main herbs, which have been used in the Orient for nearly 2000 years for a variety of GI symptoms including diarrhea and nausea/vomiting. Extensive pre-clinical research has been done with Chinese herbal medicine, and studies have documented significant anticancer activity in combination with various cytotoxic agents including Irinotecan, which is a semi-synthetic derivative of the natural alkaloid camptothecin and belongs to the class of topoisomerase I inhibitors. Irinotecan has been evaluated extensively as a single agent as well as in combination with other cytotoxic agents in several schedules. We recently completed a phase I study of irinotecan using the every-2-week schedule in combination with varying doses of KD018. Based on this phase I study, the dose of irinotecan that will be used in this study is 215 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed metastatic colorectal cancer (mCRC), who have received and/or progressed on a prior oxaliplatin-based chemotherapy regimen.
2. Patients must have been off of chemotherapy for at least 4 weeks prior to signing the informed consent/start of screening.
3. Patients with wild-type or mutant KRAS mCRC.
4. At least one measurable lesion by RECIST 1.1.
5. ECOG PS Performance Status 0-2.
6. Must be >/=18 years of age.
7. Expected survival of at least 6 months.
8. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods. Pregnant and nursing patients are excluded because the effects of the combination of KD018 and irinotecan on a fetus or nursing child are unknown.
9. Must be able and willing to give written informed consent.
10. Patients must have the following clinical laboratory values:

    1. ANC count >/= 1,500/ mm3.
    2. Platelets >/= 100,000/ mm3.
    3. Hemoglobin >/= 9 gm/dL (may be corrected by transfusion).
11. Evidence of adequate hepatic function, Bilirubin < 1.5 x upper limit of normal (ULN) AST </= 2.5 x ULN or ALT </= 2.5 x ULN (Note, if both AST and ALT are done, both must be </= 2.5 x ULN) OR AST </= 5.0 x ULN or ALT </= 5.0 x ULN is acceptable if liver has tumor involvement. (Note, if both AST and ALT are done, both must be </= 5.0 x ULN)
12. Serum creatinine </=2 x ULN
13. Serum potassium within institutional limits of normal (may be corrected with potassium repletion).

Exclusion Criteria:

1. Continued treatment with bevacizumab with documented evidence of disease progression on a bevacizumab-containing regimen.
2. Uncontrolled or symptomatic brain metastasis.
3. Serious concomitant systemic disorders (e.g., active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
4. Unwilling or unable to follow protocol requirements or to give informed consent.
5. No treatment with cytotoxic or biologic agents within the 4 weeks prior to beginning treatment on this study (6 weeks for mitomycin or nitrosoureas). At least 4 weeks must have elapsed from any prior surgery, radiation, hormonal or other drug therapy for their cancer.
6. Known HIV positivity, as safety in this patient population has not been assessed.
7. Presence of metastatic disease that, in the opinion of the investigator, would require palliative treatment within 4 weeks of enrollment.
8. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.
9. Pregnant or breast-feeding women.
10. Men and women of childbearing age and potential, who are not willing to use effective contraception.
11. Major surgery within the previous 4 weeks.
12. Patients taking concurrent medications of any kind which are strong inducers or inhibitors of CYP3A4.
13. Patients previously treated with an irinotecan-containing regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-12; Primary Completion 2016-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chu, MD, Principal Investigator — Hillman Cancer Center
Locations (2):
- United States (2):
  - Yale University Comprehensive Cancer Center, New Haven, Connecticut
  - Hillman CancerCenters, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Lam W, Bussom S, Guan F, Jiang Z, Zhang W, Gullen EA, Liu SH, Cheng YC. The four-herb Chinese medicine PHY906 reduces chemotherapy-induced gastrointestinal toxicity. Sci Transl Med. 2010 Aug 18;2(45):45ra59. doi: 10.1126/scitranslmed.3001270. PMID 20720216

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan+ KD018: KD018: Traditional Chinese Medicine formulation administered orally twice a day for 4 days on days 1-4 every 2 weeks from the second cycle, at a dose of 1,800 mg, twice a day.
  Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
- Irinotecan + Placebo: Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
  Placebo: Placebo capsules will be administered orally twice a day for 4 days on days 1-4 every 2 weeks.
Period: Overall Study
Arm/Group | Irinotecan+ KD018 | Irinotecan + Placebo
Started | 17 | 16
Completed | 16 | 15
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan+ KD018 | Irinotecan + Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (12.4) | 57.6 (12.7) | 61.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 14 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Grade 2-4 Toxicities
Description: The proportion of participants with a toxicity grade greater than or equal to grade 2, per NCI CTCAE 4.0. Toxicity is defined as any adverse event (AE) at least probably related to treatment occurring with 90 days of the beginning of treatment. The worst grade of AE at least probably related to treatment was determined for each participant.
Time Frame: Up to 3 months after start of study treatment
Population: Participants that received at least 3 months of study treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm A - Irinotecan + KD018: KD018: Traditional Chinese Medicine formulation administered orally twice a day for 4 days on days 1-4 every 2 weeks from the second cycle, at a dose of 1,800 mg, twice a day.
  Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
- Arm B - Irinotecan + Placebo: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
  Placebo: Placebo capsules will be administered orally twice a day for 4 days on days 1-4 every 2 weeks.
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 16 | 15
proportion of participants | 0.63 [0.35 to 0.85] | 0.40 [0.16 to 0.68]

2. Secondary Outcome: Overall Response (OR)
Description: Number of participants who experienced a best response of Partial Response (PR) or Stable Disease (SD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1), PR is >=30% decrease in the sum of the longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameter.
Time Frame: Up to 36 months
Population: Participants evaluable for response.
Measure: Number; unit: participants
Groups:
- Arm A - Irinotecan + KD018: Traditional Chinese Medicine formulation administered orally twice a day for 4 days on days 1-4 every 2 weeks from the second cycle, at a dose of 1,800 mg, twice a day.
  Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
- Arm B - Irinotecan + Placebo: Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m²..
  Placebo: Placebo capsules will be administered orally twice a day for 4 days on days 1-4 every 2 weeks.
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 12
participants | 7 | 10

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Median number of days and after the treatment participants remained alive without worsening disease.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 450 days
Population: Patients that were evaluable for response and survival data were obtainable.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Arm B - Irinotecan + Placebo: Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
  Placebo: Placebo capsules will be administered orally twice a day for 4 days on days 1-4 every 2 weeks.
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 12 | 14
Days | 122 [106 to NA] — Statistically Not Reached. | 104 [52 to 242]

4. Secondary Outcome: Overall Survival (OS)
Description: Median number of days from the start of treatment that study participants remained alive.
Time Frame: Up to 900 days
Population: All participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 16 | 15
Days | 291 [174 to NA] — Statistically Not Reached | 482 [308 to NA] — Statistically Not Reached

5. Secondary Outcome: Clinical Response (CR)
Description: Number of patients that experienced Progressed Disease, Stable Disease or Partial Response per RECIST 1.1. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters, and Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 36 months
Population: Participants that were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 12
participants
  Progressed Disease | 7 | 2
  Stable Disease | 5 | 9
  Partial Response | 2 | 1

6. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy (Diarrhea) FACIT-D Total Score
Description: The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System is a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness. The Functional Assessment of Chronic Illness Therapy (Diarrhea), the FACIT-D, contains 11 items which address concerns related to treatment-related diarrhea. Responses are on a Likert scale and range from 0 = "Not at all" to 4 = "Very Much". Thus, total scores can range from 0 to 44. Higher scores relate to better functioning.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACIT-D during any single treatment cycle (every 2 weeks).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 12 | 13
score on a scale
  Cycle 0 | 40.09 [36.02 to 44.16] | 39.77 [36.98 to 42.56]
  Cycle 1 | 37.66 [34.37 to 40.95] | 35.55 [30.98 to 40.12]
  Cycle 2 | 34.78 [28.57 to 40.98] | 37.78 [33.09 to 42.47]
  Cycle 3 | 37.75 [32.64 to 42.86] | 35.65 [29.48 to 41.82]
  Cycle 4 | 35.62 [30.10 to 41.15] | 35.71 [29.89 to 41.53]
  Cycle 5 | 37.09 [29.93 to 44.24] | 31.25 [25.53 to 36.97]
  Cycle 6 | 36.54 [29.52 to 43.57] | 30.38 [19.30 to 41.47]
  Cycle 7 | 38.60 [31.49 to 45.71] | 29.33 [19.06 to 39.61]
  Cycle 8 | 38.50 [23.10 to 53.90] | 28.20 [18.14 to 38.26]
  Cycle 9 | 35.67 [16.69 to 54.64] | 32.50 [0.73 to 64.27]
  Cycle 10 | 30.00 [4.59 to 55.41] | 31.50 [-25.68 to 88.68]

7. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D - PWB: Physical Well-Being
Description: The Functional Assessment of Chronic Illness Therapy FACIT-D - PWB: Physical Well-Being is a 7-item subscale score of the total FACIT-D self-assessment that measures a patient's physical well-being. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-28. Higher scores related to better physical well-being.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-Fatigue FS during any single treatment cycle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  Cycle 0 | 23.18 [21.09 to 25.27] | 21.79 [18.14 to 25.43]
  Cycle 1 | 21.69 [17.70 to 25.68] | 22.00 [18.64 to 25.36]
  Cycle 2 | 22.00 [18.27 to 25.73] | 22.21 [18.64 to 25.78]
  Cycle 3 | 24.26 [22.40 to 26.12] | 21.30 [17.18 to 25.42]
  Cycle 4 | 22.67 [20.12 to 25.22] | 23.09 [20.62 to 25.56]
  Cycle 5 | 23.62 [20.95 to 26.30] | 21.88 [17.08 to 26.67]
  Cycle 6 | 23.50 [21.09 to 25.91] | 20.00 [14.37 to 25.22]
  Cycle 7 | 22.14 [19.67 to 24.61] | 20.83 [16.31 to 25.36]
  Cycle 8 | 22.67 [19.37 to 25.96] | 17.40 [11.81 to 22.99]
  Cycle 9 | 22.00 [15.64 to 28.36] | 22.50 [-9.27 to 54.27]
  Cycle 10 | 23.33 [10.83 to 35.84] | 23.50 [17.15 to 29.85]

8. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D EWB: Emotional Well-Being
Description: The Functional Assessment of Chronic Illness Therapy FACIT-D Emotional Well-Being (EWB) is a 6-item subscale score of the total FACIT-D self-assessment that measures a patient's emotional well-being. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-24. Higher scores related to better emotional well-being.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-Fatigue FS during any single treatment cycle (every 2 weeks).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  Cycle 0 | 19.85 [17.87 to 21.82] | 16.43 [13.48 to 19.38]
  Cycle 1 | 18.00 [15.19 to 20.81] | 16.43 [13.33 to 19.53]
  Cycle 2 | 19.96 [17.36 to 22.55] | 17.30 [14.06 to 20.54]
  Cycle 3 | 20.11 [17.52 to 22.70] | 17.76 [14.11 to 21.41]
  Cycle 4 | 19.33 [16.76 to 21.91] | 19.55 [17.39 to 21.70]
  Cycle 5 | 20.38 [17.81 to 22.94] | 18.75 [15.22 to 22.28]
  Cycle 6 | 19.88 [17.53 to 22.22] | 17.20 [11.35 to 23.05]
  Cycle 7 | 20.57 [18.25 to 22.89] | 17.80 [12.95 to 22.65]
  Cycle 8 | 20.33 [17.88 to 22.79] | 15.50 [6.00 to 25.00]
  Cycle 9 | 21.25 [16.87 to 25.63] | 21.00 [-4.41 to 46.41]
  Cycle 10 | 22.00 [17.03 to 26.97] | 20.30 [3.78 to 36.82]

9. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D SWB: Social Well-Being
Description: The Functional Assessment of Chronic Illness Therapy FACIT-D Social Well-Being (SWB) is a 7-item subset score of the total FACIT-D self-assessment that measures a patient's social well-being. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-28. Higher scores related to better social well-being.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-Fatigue FS during any single treatment cycle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  Cycle 0 | 25.85 [24.74 to 26.96] | 23.91 [20.52 to 27.29]
  Cycle 1 | 21.46 [17.01 to 25.92] | 24.33 [21.30 to 27.36]
  Cycle 2 | 20.74 [14.07 to 27.41] | 25.60 [23.70 to 27.50]
  Cycle 3 | 25.09 [22.16 to 28.03] | 25.33 [23.74 to 26.91]
  Cycle 4 | 23.43 [20.17 to 26.68] | 24.60 [21.23 to 27.97]
  Cycle 5 | 25.07 [21.71 to 28.44] | 24.29 [19.09 to 29.49]
  Cycle 6 | 22.19 [15.33 to 29.04] | 23.60 [21.90 to 24.21]
  Cycle 7 | 25.83 [21.76 to 29.91] | 22.89 [19.05 to 26.73]
  Cycle 8 | 24.22 [19.58 to 28.87] | 21.63 [15.45 to 27.82]
  Cycle 9 | 25.67 [20.42 to 30.92] | 23.00 [-2.41 to 48.41]
  Cycle 10 | 24.94 [14.21 to 35.68] | 23.50 [-8.27 to 55.27]

10. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D FWB: Functional Well-Being
Description: The Functional Assessment of Chronic Illness Therapy FACIT-D Functional Well-Being (FWB) is a 7-item subscale of the FACIT-D that measures a patient's functional well-being. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-28. Higher scores related to better family well-being.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-Fatigue FS during any single treatment cycle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  Cycle 0 | 19.85 [16.48 to 23.21] | 18.07 [14.44 to 21.70]
  Cycle 1 | 18.89 [14.62 to 23.17] | 17.21 [13.84 to 20.59]
  Cycle 2 | 19.78 [15.43 to 24.97] | 20.20 [14.46 to 25.10]
  Cycle 3 | 20.11 [15.59 to 24.63] | 19.32 [14.33 to 24.30]
  Cycle 4 | 19.44 [15.47 to 23.42] | 19.09 [14.86 to 23.32]
  Cycle 5 | 19.77 [16.09 to 23.46] | 20.50 [10.56 to 30.44]
  Cycle 6 | 19.62 [15.48 to 23.77] | 17.00 [10.31 to 23.69]
  Cycle 7 | 19.00 [12.98 to 25.02] | 16.40 [10.74 to 22.06]
  Cycle 8 | 19.83 [14.85 to 24.82] | 17.00 [7.19 to 26.81]
  Cycle 9 | 22.58 [7.19 to 26.81] | 20.50 [14.85 to 24.82]
  Cycle 10 | 21.00 [-35.68 to 78.68] | 21.50 [2.25 to 39.75]

11. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D FACTG: FACT-G Total Score (PWB+SWB+EWB+FWB)
Description: The FACIT-D FACTG: FACT-G Total Score is a total of PWB (Physical Well-Being)+SWB (Social Well-Being)+EWB (Emotional Well-Being)+FWB (Functional Well-Being) subset scores. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-108. Higher scores indicate greater well-being.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-G during any single treatment cycle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Arm A - Irinotecan+ KD018: KD018: Traditional Chinese Medicine formulation administered orally twice a day for 4 days on days 1-4 every 2 weeks from the second cycle, at a dose of 1,800 mg, twice a day.
  Irinotecan: Irinotecan will be administered intravenously once every 2 weeks from the first cycle, at a dose of 215 mg/m².
Arm/Group | Arm A - Irinotecan+ KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 13 | 14
score on a scale
  Cycle 0 | 88.72 [82.18 to 95.26] | 80.19 [68.66 to 91.73]
  Cycle 1 | 80.05 [68.46 to 91.64] | 79.98 [69.37 to 90.58]
  Cycle 2 | 82.47 [69.52 to 95.42] | 84.99 [72.48 to 97.51]
  Cycle 3 | 89.57 [79.78 to 99.37] | 83.70 [70.54 to 96.86]
  Cycle 4 | 84.87 [75.61 to 94.13] | 86.33 [76.32 to 96.33]
  Cycle 5 | 88.85 [78.33 to 99.36] | 85.42 [64.40 to 106.44]
  Cycle 6 | 85.19 [73.99 to 96.38] | 79.07 [65.44 to 92.70]
  Cycle 7 | 87.55 [75.96 to 99.13] | 76.43 [60.23 to 92.62]
  Cycle 8 | 87.06 [74.44 to 99.67] | 74.79 [48.58 to 101.00]
  Cycle 9 | 91.50 [73.24 to 109.76] | 87.00 [-65.47 to 239.47]
  Cycle 10 | 91.28 [53.15 to 129.40] | 88.80 [-23.01 to 200.61]

12. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-Fatigue FS: Fatigue Score
Description: The Functional Assessment of Chronic Illness Therapy FACIT-Fatigue FS: Fatigue Score is a 13 -item self-reporting assessment that measures fatigue related to their illness. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score ranges from 0-52. Higher scores indicate better functioning.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACT-Fatigue FS during any single treatment cycle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 13 | 12
score on a scale
  Cycle 0 | 41.39 [36.50 to 46.28] | 36.17 [28.42 to 43.91]
  Cycle 1 | 36.09 [26.22 to 45.96] | 36.67 [30.36 to 42.97]
  Cycle 2 | 38.80 [32.68 to 44.92] | 38.45 [30.44 to 46.47]
  Cycle 3 | 41.67 [36.57 to 46.77] | 36.22 [27.19 to 45.26]
  Cycle 4 | 40.22 [36.18 to 44.27] | 38.56 [30.64 to 46.47]
  Cycle 5 | 40.25 [36.02 to 44.48] | 39.75 [23.77 to 55.73]
  Cycle 6 | 41.53 [36.03 to 47.03] | 30.72 [20.11 to 41.33]
  Cycle 7 | 41.33 [34.67 to 47.99] | 33.33 [22.74 to 43.93]
  Cycle 8 | 40.78 [28.92 to 52.65] | 30.20 [14.96 to 45.44]
  Cycle 9 | 40.25 [29.59 to 50.91] | 33.33 [-1.47 to 68.14]
  Cycle 10 | 41.50 [30.14 to 52.86] | 40.00 [-36.24 to 116.24]

13. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy FACIT-D TOI: Trial Outcome Index
Description: The Functional Assessment of Chronic Illness Therapy FACIT-D TOI: Trial Outcome Index. is the sum of the Physical Well-Being (PWB), Functional Well-Being (FWB), and "additional concerns" subscales of the FACIT-D. The TOI is an efficient summary index of physical/functional outcomes. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System is a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness. Individual responses are scale and range from 0 = "Not at all" to 4 = "Very Much". The total score can range from 0-100. Higher scores relate to better functioning.
Time Frame: Up to 36 months
Population: Maximum number of participants that completed the FACIT-D during any single treatment cycle (every 2 weeks).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A - Irinotecan+ KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 13 | 12
score on a scale
  Cycle 0 | 82.03 [75.36 to 88.70] | 79.23 [71.42 to 87.04]
  Cycle 1 | 78.01 [68.39 to 87.63] | 75.17 [66.46 to 83.89]
  Cycle 2 | 76.56 [62.84 to 90.27] | 82.42 [72.85 to 91.98]
  Cycle 3 | 81.88 [71.97 to 91.78] | 76.27 [62.73 to 89.80]
  Cycle 4 | 77.12 [68.15 to 86.10] | 79.11 [67.99 to 90.23]
  Cycle 5 | 80.40 [67.97 to 92.82] | 73.62 [56.42 to 90.83]
  Cycle 6 | 79.11 [68.09 to 90.14] | 66.46 [47.02 to 85.90]
  Cycle 7 | 82.00 [67.33 to 96.67] | 65.40 [47.27 to 83.53]
  Cycle 8 | 81.25 [55.74 to 106.76] | 61.50 [33.62 to 89.38]
  Cycle 9 | 80.44 [38.37 to 122.52] | 75.50 [-57.92 to 208.92]
  Cycle 10 | 68.50 [-1.38 to 138.38] | 76.50 [-44.21 to 197.21]

14. Secondary Outcome: Metabolites and Cytokine Scoring for Prediction of Time to Disease Progression
Description: Number of patients with metabolites in their blood samples with a score less than 4.8 and greater than 4.8. A Cox Proportional Hazard Regression Analysis was fitted using survival time, status to the cytokines and metabolites as covariates. The analysis computes beta coefficients (hazard ratios) for each cytokine/metabolite. Scores higher than a threshold value of 4.8 were associated with higher overall survival than patients who scored less than 4.8.
Time Frame: Up to 36 months
Population: Patients that received study treatment.
Measure: Number; unit: participants
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 8 | 9
participants
  Scores < 4.8 (two metabolites) | 3 | 3
  Scores > 4.8 (two metabolites) | 5 | 6
  Scores < 4.8 (one metabolite+two cytokine) | 2 | 4
  Scores > 4.8 (one metabolite+two cytokine) | 6 | 5

15. Secondary Outcome: Uridine Diphosphate Glucuronosyltransferase (UGT) 1A1 Alleles
Description: The number of patients with specific polymorphisms of UGT1A1 using genotype analysis of peripheral blood sample. UGT1A1*1 is the wild-type allele associated with normal enzyme activity. Patients with genotypic status of 7/7 are at an increased risk of neutropenia following intravenous irinotecan therapy.
Time Frame: From 30 minutes prior to irinotecan infusion through to Immediately after irinotecan infusion, up to 8 weeks
Population: Patients who completed at least (3) treatment cycles.
Measure: Number; unit: number of participants
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 12
number of participants
  genotype 5/6 | 0 | 1
  genotype 6/6 | 4 | 4
  genotype 6/7 | 5 | 4
  genotype 7/7 | 0 | 0

16. Secondary Outcome: Circulating Tumor DNA - Percentage of Patients With DNA Mutations
Description: Percentage of patients with Braf, Kras, Nras, PIK3CA and PTEN mutations associated with tumor detected in the circulating DNA of plasma, before treatment.
Time Frame: Baseline - prior to treatment
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 12
percentage of participants
  Braf mutation | 22 | 22
  Kras mutation | 66 | 44
  Nras mutation | 11 | 0
  PIK3CA mutation | 22 | 55
  PTEN mutation | 11 | 11

17. Secondary Outcome: Circulating Tumor DNA - Percentage of Patients With DNA Mutations
Description: as for outcome 16
Time Frame: End of treatment - up to 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Irinotecan+ KD018 | Arm B - Irinotecan + Placebo
Number analyzed (Participants) | 14 | 12
percentage of participants
  Braf mutation | 0 | 22
  Kras mutation | 33 | 44
  Nras mutation | 11 | 11
  PIK3CA mutation | 22 | 0
  PTEN mutation | 11 | 11

ADVERSE EVENTS:
Arm/Group | Arm A - Irinotecan + KD018 | Arm B - Irinotecan + Placebo
Serious Adverse Events (participants affected / at risk) | 3/16 | 4/15
Other Adverse Events (participants affected / at risk) | 11/16 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Irinotecan + KD018 (N=16) | Arm B - Irinotecan + Placebo (N=15)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Blood bilirubin increased (Investigations) | 1 (7) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
INR increased (Investigations) | 1 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (8) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
White blood cell decreased (Investigations) | 2 (4) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Irinotecan + KD018 (N=16) | Arm B - Irinotecan + Placebo (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (12)
Alanine aminotransferase increased (Investigations) | 3 (14) | 3 (20)
Alkaline phosphatase increased (Investigations) | 3 (8) | 4 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (20) | 5 (16)
Anemia (Blood and lymphatic system disorders) | 6 (36) | 7 (48)
Anorexia (Metabolism and nutrition disorders) | 1 (4) | 3 (9)
Anxiety (Psychiatric disorders) | 3 (6) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 4 (14) | 5 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (8)
Bloating (Gastrointestinal disorders) | 1 (4) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (11) | 2 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 1 (2) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (12) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Creatinine increased (Investigations) | 1 (4) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Depression (Psychiatric disorders) | 2 (4) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 10 (70) | 10 (77)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (4)
Dysarthria (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 1 (2)
Edema limbs (General disorders) | 2 (4) | 0 (0)
Edema trunk (General disorders) | 1 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 11 (36) | 9 (23)
Fecal incontinence (Gastrointestinal disorders) | 1 (2) | 1 (2)
Fever (General disorders) | 2 (4) | 1 (2)
Flatulence (Gastrointestinal disorders) | 3 (12) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (34) | 4 (10)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (10) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (4)
Hallucinations (Psychiatric disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (4)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (18) | 1 (2)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (16) | 2 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hypertension (Vascular disorders) | 2 (4) | 1 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 2 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (26) | 5 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (18) | 4 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8) | 3 (14)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (26) | 4 (10)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 4 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (36) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
INR increased (Investigations) | 2 (6) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (2)
Investigations - Other, specify (Investigations) | 2 (6) | 1 (4)
Localized edema (General disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (62) | 1 (6)
Lymphocyte count increased (Investigations) | 2 (6) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Nausea (Gastrointestinal disorders) | 11 (42) | 7 (39)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (8) | 1 (2)
Neutrophil count decreased (Investigations) | 8 (48) | 7 (22)
Pain (General disorders) | 4 (14) | 2 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4) | 1 (1)
Platelet count decreased (Investigations) | 2 (6) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 2 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 2 (4)
Restlessness (Psychiatric disorders) | 1 (2) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (12) | 7 (27)
Weight loss (Investigations) | 3 (8) | 2 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
White blood cell decreased (Investigations) | 10 (72) | 5 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes